CLINICAL TRIAL: NCT03023917
Title: The Study on Umbilical Cord Milking to Prevent and Decrease the Severity of Anemia in preterms--a Multi-center Randomized Controlled Trial
Brief Title: The Study on Umbilical Cord Milking to Prevent and Decrease the Severity of Anemia in Preterms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai First Maternity and Infant Hospital (Other); Yangpu District Central Hospital Affiliated to Tongji University (Other)
Responsible Party: Principal Investigator, Lijuan Xie, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XH-16-050
Record Dates: First submitted 2017-01-03; First posted 2017-01-18 (Estimated); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Anemia
Keywords: umbilical cord milking;anemia;placental transfusion
MeSH Terms: conditions — Anemia | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- umbilical cord clamping immediately (Active Comparator): Umbilical cord was clamped immediately, or as close as possible, after delivery of the infant's shoulders. (This was standard practice in the study hospital, thus it served as the "control" group).
  Interventions: Procedure: umbilical cord clamping immediately
- umbilical cord milking (Experimental): preterm baby were placed at or below level of the placenta and about 25cm of the umbilical cord was vigorously milked towards the umbilicus two to three times before clamping the cord. The milking speed was about 25cm/2 seconds
  Interventions: Procedure: umbilical cord milking

INTERVENTIONS:
Procedure: umbilical cord milking — Infants were placed at or below level of the placenta and about 25cm of the umbilical cord was vigorously milked towards the umbilicus two to three times before clamping the cord. The milking speed was about 25cm/2 seconds
  Arms: umbilical cord milking
Procedure: umbilical cord clamping immediately — umbilical cord was cut immediately after birth
  Arms: umbilical cord clamping immediately

SUMMARY:
The overall objective of the present study is to examine the effects of umbilical cord milking at birth in preterm infants to prevent and decrease anemia using a multi-center prospective randomized controlled trial comparing immediate cord clamping (standard at present) with umbilical cord milking.

DETAILED DESCRIPTION:
Anemia is a significant problem for pre-term infants and a major risk factor for preterm babies mortality and morbidity in neonatal intensive care unit(NICU). the majority of pre-term babies will require one or more blood transfusions during in NICU. Blood transfusion is a safe procedure but like all therapeutic interventions has risks associated with it and effort is made to reduce the number of transfusions that infants require during their stay on the neonatal unit.

Delayed cord clamping has a beneficial effect on prevention of anemia in later infancy because of increased iron stores at birth. However there are controversies in incorporating delayed cord clamping practice in the management of third stage of labour globally. Concerning about the need for urgent resuscitation and temperature management, attendants encouraged to clamp the umbilical cord immediately so that post-natal resuscitation and care can start as soon as possible.However,umbilical cord milking allows for swift intervention and resuscitation and attention to thermal care and should take less than 10 seconds to complete.

The specific aim of this study is to investigate the effects of umbilical cord milking on preventing and decreasing anemia in very pre-term infants.

Primary Outcomes:

Hemoglobin (Hb), Hematocrit (Hct) and serum iron levels at birth, at 1 week,at 2 weeks of age.

Secondary Outcomes:

* Hemoglobin,hematocrit levels at 6 months of age.
* Anemia at 1 week of life and 6 months follow-up, defined as hemoglobin levels below the respective cutoffs.
* number of blood transfusions until 3 months corrected gestational age (CGA).
* short term clinical profile of neonates like jaundice, polycythemia etc.
* preterm infant complications such as lung function as assessed by oxygen dependency at 36 weeks corrected gestational age (CGA), and cardiovascular function as assessed by the need for volume expansion, inotropes, or clinically suspected patent ductus arteriosus(PDA )requiring intervention prior to discharge home,incidence of intraventricular hemorrhage and late-onset sepsis,etc.

ELIGIBILITY:
Inclusion Criteria:

* Women in labour or with a plan for delivery at a gestational age less than 34 weeks gestation.
* Singleton pregnancy
* informed consent was obtained from the parent

Exclusion Criteria:

* Multiple gestation
* Diagnosis of any of the following in the current pregnancy: hemorrhage requiring clinic/hospital admission, placental abnormalities, fetal anomalies, Down's syndrome of the fetus,anemia
* Diagnosis of pre-eclampsia or eclampsia in current or previous pregnancies
* Diagnosis at any time for the mother of any of the following: serious Diabetes, serious hypertension, chronic renal disease
* Infant with major congenital malformation
* Infant with blood disease
* Unwilling to return for follow-up study visits at the hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
concentrations of Hemoglobin (Hb) | 48 hours after birth
concentrations of Hematocrit(Hct) | 48 hours after birth
serum ferritin level | 48 hours after birth

SECONDARY OUTCOMES:
Hyperbilirubinemia requiring phototherapy | during first 2 weeks of age
  Hyperbilirubinemia requiring phototherapy (as per routine unit practice)
incidence and numbers of blood transfusions | until 3 months corrected gestational age
Length of admission | Birth to discharge, expected average of 30 days
complication | Birth to discharge, expected average of 30 days
  composite of bronchopulmonary dysplasia , Necrotizing Enterocolitis , grade 3 or 4 intraventricular hemorrhage or periventricular leukomalacia , or death prior to discharge home

CONTACTS AND LOCATIONS:
Overall Officials: guangyu chen, Study Chair — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No